CLINICAL TRIAL: NCT06825533
Title: The Prevalence of Prediabetes in Primary Care Medicine in Tunisia. a National Descriptive Cross-Sectional Study
Brief Title: The Prevalence of Prediabetes in Primary Care Medicine in Tunisia
Acronym: TUN-PREDIAB
Status: Not yet recruiting | Type: Observational
Sponsor: Dacima Consulting (Other)
Collaborators: Société Tunisienne de Médecine Générale et de Médecine de Famille (Unknown)
Responsible Party: Sponsor
Other Study IDs: DAC-016-TUN-PREDIAB
Record Dates: First submitted 2025-02-09; First posted 2025-02-13 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Prediabetes
Keywords: Prediabetes; STMGF; Survey
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Fasting blood sugar level — Assess the level of Blood sugar level in fasting conditions at inclusion
Diagnostic Test: Glycated hemoglobin — Assess the level of glycated hemoglobin at inclusion

SUMMARY:
The study is national, observational and cross-sectional and aims to estimate the prevalence of prediabetes in primary care in Tunisia.

DETAILED DESCRIPTION:
TN-PREDIAB is a Tunisian, descriptive, non-interventional, multicenter and cross-sectional clinical study performed in primary care facilities, of both public and private sectors. The study will screen ambulatory patients for at least 4 months to estimate the prevalence of prediabetes among enrolled subjects.

The objectives of the study are:

* Primary objective: to estimate the overall prevalence of prediabetes among Tunisian population
* Secondary objective:
* Describe the clinical and epidemiological profile of prediabetic subjects
* Describe nutritional factors associated with prediabetes

A Scientific Committee validates the scientific writing, a Steering Committee supervises the clinical operations of the project.

Collected data are managed by the DACIMA Clinical Suite®, the electronic data capture platform which complies with the FDA 21 CFR part 11 requirements (Food and Drug Administration 21 Code of Federal Regulations part 11), the HIPAA specifications (Health Insurance Portability and Accountability Act), and the ICH standards (International Conference on Harmonisation).

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory patient consulting in primary care in a public or private structure

Exclusion Criteria:

* Known diabetes
* Concomitant medication that may influence blood sugar (corticosteroids, metformin, GLP1 analogues, SGLT2 inhibitor)
* Severe, acute or chronic comorbidity (end-stage renal failure, severe liver disease, heart failure)
* Severe anemia
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ambulatory patient consulting in primary care in a public or private structure, without patent diabetes
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2025-04-21 (Estimated); Primary Completion 2025-08-21 (Estimated); Study Completion 2025-08-21 (Estimated)

PRIMARY OUTCOMES:
Prediabetes | At inclusion
  Percentage of prediabetic patients discovered at inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Haithem Ben Haj Salah, MD, Study Chair — Société Tunisienne de Médecine Générale et de Médecine de Famille; Habib Jerbi, MD, Study Chair — Société Tunisienne de Médecine Générale et de Médecine de Famille

IPD SHARING:
Plan to Share IPD: No